CLINICAL TRIAL: NCT02192554
Title: A 2-Month, Observational, Rollover Trial to Evaluate the Safety of Subjects With Agitation Associated With Dementia of the Alzheimer's Type Who Were Previously Treated With Brexpiprazole (OPC 34712) or Placebo in a Phase 3, Double-blind Trial
Brief Title: Safety Follow-up Study for Subjects With Agitation Associated With Dementia of the Alzheimer's Type Who Previously Participated in a Double-blind Trial of Brexpiprazole or Placebo
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 331-13-211
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Agitation Associated With Alzheimer's Disease; Alzheimer's Type; Mental Disorder; Nervous System Diseases
Keywords: OPC-34712; brexpiprazole; Dementia; Alzheimer's Disease; Cognitive Disorders; Memory; Agitation
MeSH Terms: conditions — Mental Disorders; Nervous System Diseases; Dementia; Alzheimer Disease; Cognitive Dysfunction; Psychomotor Agitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To follow-up on the safety of subjects who were previously treated in a double-blind trial of brexpiprazole.

DETAILED DESCRIPTION:
Behavioral symptoms, such as agitation, are core features in subjects with Alzheimer's disease and related dementias, and develop in the majority of dementia subjects. The presence of agitation in subjects with Alzheimer's disease places a significant burden not only on subjects and their caregivers but also on the healthcare system.

This is a trial designed to assess the ongoing safety of subjects with agitation associated with dementia of the Alzheimer's type after completing a 12-week double-blind trial of brexpiprazole or placebo; drug and placebo are discontinued prior to subjects enrolling in the safety follow-up trial. The trial consists of a continuous 2 month observation period. The trial population will include male and female subjects with a diagnosis of probable Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* The investigator must assess the capacity of the subject to provide informed consent prior to enrollment and throughout the trial.
* Male and female subjects who completed both the 12-week double-blind treatment period and the 30-day safety follow-up visit of the previous brexpiprazole trial.
* Subject has an identified caregiver who is usually assigned to care for the subject on a regular basis, has sufficient contact to describe the subject's symptoms, and has direct observation of the subject's behavior.
* Subject is able to comply with the protocol requirements.

Exclusion Criterion:

* Subjects who, in the opinion of the investigator, medical monitor, or sponsor should not participate in the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects must have completed a previous double-blind trial of brexpiprazole or placebo; neither drug or placebo will be administered in the trial
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Baseline to Month 2/Early Termination
Mini-Mental State Examination (MMSE) score | Baseline to Month 2/Early Termination

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kohegyi, MD, MS, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (68):
- United States (24):
  - Tuscaloosa, Alabama
  - Costa Mesa, California
  - Lakewood, California
  - Orange, California
  - Redlands, California
  - Bradenton, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Miami Springs, Florida
  - North Miami, Florida
  - Orange City, Florida
  - Sarasota, Florida
  - Atlanta, Georgia
  - Suwanee, Georgia
  - Quincy, Massachusetts
  - St Louis, Missouri
  - Toms River, New Jersey
  - Brooklyn, New York
  - New Hyde Park, New York
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Dallas, Texas
  - Waukesha, Wisconsin
- Bulgaria (6):
  - Burgas
  - Kardzhali
  - Rousse
  - Sofia
  - Varna
  - Veliko Tarnovo
- Canada (2):
  - Penticton, British Columbia
  - Kentville, Nova Scotia
- Zagreb, Croatia
- France (4):
  - Bourg N Bresse
  - Douai
  - Élancourt
  - Toulouse
- Germany (5):
  - Mittweida, Saxony
  - Berlin
  - Bochum
  - Cologne
  - Westerstede
- Russia (5):
  - Saint Petersburg
  - Samara
  - Saratov
  - Tonnelniy
  - Yekaterinburg
- Serbia (6):
  - Belgrade
  - Kovin
  - Kragujevac
  - Niš
  - Novi Kneževac
  - Novi Sad
- Slovenia (3):
  - Ljubljana
  - Maribor
  - Šempeter pri Gorici
- Spain (4):
  - Pamplona
  - Salamanca
  - Valencia
  - Zamora
- Ukraine (7):
  - Kharkiv
  - Kherson
  - Kiev
  - Lviv
  - Odesa
  - Poltava
  - Vinnytsia
- Torpoint, United Kingdom